CLINICAL TRIAL: NCT04147546
Title: Operational Feasibility, Impact of Additional Screening Using Highly-sensitives RDTs Combined With High Coverage of IPTp on Placental Malaria and Low Birth Weight
Brief Title: Additional Screening With Sensitives RDTs and Malaria
Acronym: ASSERMalaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NCT04147546
Record Dates: First submitted 2019-10-14; First posted 2019-11-01 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Plasmodium Falciparum Malaria; Malaria Diagnosis
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): A full course of dihydroartemisinin-piperaquine (DP) over 3 days. The first dose of DP will be administered under direct observation at the antenatal care clinic (ANC) and the subsequent doses of the intervention in days 2 and 3 will be taken unsupervised at home.
  At each ANC visit, study nurses will perform an HS-RDT for participants in this arm. Reminders will be sent in this group in order to improve IPTp-SP uptake
  Interventions: Diagnostic Test: Additional screening using ultra sensitive RDTs; Drug: Dihydroartemisinin-piperaquin; Other: Reminders
- Control arm (No Intervention): A full course of artemether-lumefantrine (AL) over 3 days. The first dose of AL will be administered under direct observation at the antenatal care clinic (ANC) and the subsequent doses of the intervention in days 2 and 3 will be taken unsupervised at home.
  At each ANC visit, study nurses will perform a conventional RDT for participants in this arm if the participant have symptoms suggestive of malaria. No reminder will be sent

INTERVENTIONS:
Diagnostic Test: Additional screening using ultra sensitive RDTs — At each ANC visit, study nurses will perform an HS-RDT for participants in the intervention arm
  Other Names: Malaria Ag Pf ultra-sensitive RDT
  Arms: Intervention arm
Drug: Dihydroartemisinin-piperaquin — All pregnant women with a positive HS-RDT will be treated with a full course of dihydroartemisinin-piperaquine (DP) over 3 days. The first dose of DP will be administered under direct observation at the antenatal care clinic (ANC) and the subsequent doses of the intervention in days 2 and 3 will be taken unsupervised at home
  Arms: Intervention arm
Other: Reminders — Before each scheduled ANC visit, reminders using SMS or phone call will be used. This is order to increase ANC attendance
  Arms: Intervention arm

SUMMARY:
National malaria control strategies in pregnant women relies primarily on effective case management along with the use of long lasting insecticide-treated nets (LLINs)throughout pregnancy and intermittent preventive treatment with sulfadoxine-pyrimethamine (IPTp-SP) in the second and third trimesters in malaria-endemic regions in sub-Saharan Africa (SSA). For the latter, 3 or more doses are recommended by the national malaria control program (NMCP) but available data suggests that only 19% of eligible women received this in 2016 despite observed high attendance to antenatal clinic (ANC). Adherence to IPTp may be affected by perceptions, acceptability and contextual factors that need to be understood and therefore improve the effectiveness of this health interventions. In addition, all malaria cases should be confirmed either by microscopy or using a rapid diagnostic test (RDTs) before any treatment. Despite the crucial role of RDTs in improving malaria case management SSA, many malaria cases are missed in pregnant women due to the power performance of recommended RDTs which are unable to detect very low parasitaemia. Identifying lower density infections in pregnant women by the use of highly-sensitive RDTs and clearing them with an effective ACT could improve the outcome of the pregnancy in addition to IPTp-SP.

DETAILED DESCRIPTION:
MiP remains a major public health issue in Burkina Faso, which would compromise the achievement of Sustainable Development Goals for maternal and child health (22). Malaria control program have been implemented by the Burkinabe Ministry of Health (MoH) since 2000; nevertheless, lower coverage and delays in implementation of these programs may have reduced their effectiveness.

In Burkina Faso, recommended preventions strategies for malaria imply the administration of at least 3 doses of IPTp during ANCs and before delivery (23). IPTp have been proven to have a great impact on PM, LBW and peripheral malaria infection at delivery so increasing the number of IPTp doses given is a priority. Strategies to increase the number of IPTp doses and the coverage using reminders could improve this health intervention effectiveness. This can be considered as follow up of the Cosmic study (24) recommendations.

However with increasing drug resistance, there is a progressively diminished efficacy of IPTp-SP in clearing existing infections and a shortening of the post-treatment prophylaxis period (25). Moreover, pregnant women can generally be infected with low parasites densities between ANCs compromising the outcome of the pregnancy (26). Therefore, additional screening with HS-RDTs between ANCs and treatment using ACTs with long Post-treatment prophylaxis effect in addition to IPTp-SP could have a great impact both for the mothers and their offspring's.

This proposal aims to determine the operational feasibility and the impact of additional screening with HS-RDTs and treatment with DP on placental malaria (PM) and low birth weight (LBW) in a context of IPTp-SP, in rural central Burkina Faso. The findings obtained from this study will help to assist the MoH in the implementation of the appropriate interventions in this group at risk.

Objectives

General objective

- To determine the operational feasibility and the impact of additional screening with HS-RDTs and treatment with DP on PM, LBW and peripheral malaria infection at delivery in in Burkina Faso

Specific objectives are the following:

* To determine the gain of additional screening with HS-RDTs and treatment with DP against PM, LBW and peripheral malaria infection at delivery
* To assess the determinants of the poor coverage and improve the number of IPTp doses received using phone call or SMS as a reminder

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 16 to 24 weeks at their first booking
* At least (≥) 16 years old
* Residence in the study area and intention to stay in the area for the duration of the pregnancy and for delivery
* Willing to deliver at the health facility
* Willing to provide biological samples as and when required during the study period (blood and placental biopsy)
* Ability to provide written informed consent

Exclusion Criteria:

* A history of sensitivity to sulphonamides or to any of the study drugs;
* History of known pregnancy complications or bad obstetric history such as repeated stillbirths or eclampsia;
* History or presence of major illnesses likely to influence pregnancy outcome including diabetes mellitus, severe renal or heart disease, or active tuberculosis;
* Any significant illness at the time of screening that requires hospitalization, including severe malaria;
* Intent to move out of the study catchment area before delivery or deliver at relative's home out of the catchment area.
* Prior enrolment in the study or concurrent enrolment in another study.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 340 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Placental malaria prevalence | 36 months
  The prevalence of placental malaria infection will be determined in the two arms. Placentas will be identified as not infected (no evidence of parasite or pigment); active infection (presence of parasites and pigment) and chronic infection (absence of parasites and presence of pigment)
Low birthweight prevalence | 36 months
  The prevalence of low birthweight (defined as birth weight less than 2,500 g) will be compared between the two arms.
Peripheral maternal malaria infection prevalence | 36 months
  At delivery, malaria will be diagnosed using peripheral thick smears. Parasite density will be estimated by counting the number of asexual parasites per 200 leukocytes in the thick blood film and assuming white blood cells (WBC) count of 8,000/μl

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherche en Sciences de la Santé/ Clinical Research Unit of Nanoro, Ouagadougou, Kadiogo, Burkina Faso

IPD SHARING:
Plan to Share IPD: Yes
In accordance to the EDCTP2 grant agreement, all data generated through this study will be shared in order to allow for third parties to access, mine, exploit, reproduce and disseminate, free of charge
Time Frame: At the end of the study and after all publications accepted

REFERENCES:
- [Background] Dellicour S, Tatem AJ, Guerra CA, Snow RW, ter Kuile FO. Quantifying the number of pregnancies at risk of malaria in 2007: a demographic study. PLoS Med. 2010 Jan 26;7(1):e1000221. doi: 10.1371/journal.pmed.1000221. PMID 20126256
- [Background] Desai M, ter Kuile FO, Nosten F, McGready R, Asamoa K, Brabin B, Newman RD. Epidemiology and burden of malaria in pregnancy. Lancet Infect Dis. 2007 Feb;7(2):93-104. doi: 10.1016/S1473-3099(07)70021-X. PMID 17251080
- [Background] COSMIC Consortium. Community-based Malaria Screening and Treatment for Pregnant Women Receiving Standard Intermittent Preventive Treatment With Sulfadoxine-Pyrimethamine: A Multicenter (The Gambia, Burkina Faso, and Benin) Cluster-randomized Controlled Trial. Clin Infect Dis. 2019 Feb 1;68(4):586-596. doi: 10.1093/cid/ciy522. PMID 29961848
- [Background] Radeva-Petrova D, Kayentao K, ter Kuile FO, Sinclair D, Garner P. Drugs for preventing malaria in pregnant women in endemic areas: any drug regimen versus placebo or no treatment. Cochrane Database Syst Rev. 2014 Oct 10;2014(10):CD000169. doi: 10.1002/14651858.CD000169.pub3. PMID 25300703
- [Background] van Eijk AM, Hill J, Larsen DA, Webster J, Steketee RW, Eisele TP, ter Kuile FO. Coverage of intermittent preventive treatment and insecticide-treated nets for the control of malaria during pregnancy in sub-Saharan Africa: a synthesis and meta-analysis of national survey data, 2009-11. Lancet Infect Dis. 2013 Dec;13(12):1029-42. doi: 10.1016/S1473-3099(13)70199-3. Epub 2013 Sep 18. PMID 24054085
- [Background] Gutman J, Kalilani L, Taylor S, Zhou Z, Wiegand RE, Thwai KL, Mwandama D, Khairallah C, Madanitsa M, Chaluluka E, Dzinjalamala F, Ali D, Mathanga DP, Skarbinski J, Shi YP, Meshnick S, ter Kuile FO. The A581G Mutation in the Gene Encoding Plasmodium falciparum Dihydropteroate Synthetase Reduces the Effectiveness of Sulfadoxine-Pyrimethamine Preventive Therapy in Malawian Pregnant Women. J Infect Dis. 2015 Jun 15;211(12):1997-2005. doi: 10.1093/infdis/jiu836. Epub 2015 Jan 6. PMID 25564249
- [Background] Ruizendaal E, Tahita MC, Geskus RB, Versteeg I, Scott S, d'Alessandro U, Lompo P, Derra K, Traore-Coulibaly M, de Jong MD, Schallig HDFH, Tinto H, Mens PF. Increase in the prevalence of mutations associated with sulfadoxine-pyrimethamine resistance in Plasmodium falciparum isolates collected from early to late pregnancy in Nanoro, Burkina Faso. Malar J. 2017 Apr 28;16(1):179. doi: 10.1186/s12936-017-1831-y. PMID 28454537
- [Background] Kakuru A, Jagannathan P, Muhindo MK, Natureeba P, Awori P, Nakalembe M, Opira B, Olwoch P, Ategeka J, Nayebare P, Clark TD, Feeney ME, Charlebois ED, Rizzuto G, Muehlenbachs A, Havlir DV, Kamya MR, Dorsey G. Dihydroartemisinin-Piperaquine for the Prevention of Malaria in Pregnancy. N Engl J Med. 2016 Mar 10;374(10):928-39. doi: 10.1056/NEJMoa1509150. PMID 26962728
- [Background] Hofmann NE, Gruenberg M, Nate E, Ura A, Rodriguez-Rodriguez D, Salib M, Mueller I, Smith TA, Laman M, Robinson LJ, Felger I. Assessment of ultra-sensitive malaria diagnosis versus standard molecular diagnostics for malaria elimination: an in-depth molecular community cross-sectional study. Lancet Infect Dis. 2018 Oct;18(10):1108-1116. doi: 10.1016/S1473-3099(18)30411-0. Epub 2018 Aug 28. PMID 30170986
- [Background] Das S, Jang IK, Barney B, Peck R, Rek JC, Arinaitwe E, Adrama H, Murphy M, Imwong M, Ling CL, Proux S, Haohankhunnatham W, Rist M, Seilie AM, Hanron A, Daza G, Chang M, Nakamura T, Kalnoky M, Labarre P, Murphy SC, McCarthy JS, Nosten F, Greenhouse B, Allauzen S, Domingo GJ. Performance of a High-Sensitivity Rapid Diagnostic Test for Plasmodium falciparum Malaria in Asymptomatic Individuals from Uganda and Myanmar and Naive Human Challenge Infections. Am J Trop Med Hyg. 2017 Nov;97(5):1540-1550. doi: 10.4269/ajtmh.17-0245. Epub 2017 Aug 18. PMID 28820709
- [Background] Vasquez AM, Medina AC, Tobon-Castano A, Posada M, Velez GJ, Campillo A, Gonzalez IJ, Ding X. Performance of a highly sensitive rapid diagnostic test (HS-RDT) for detecting malaria in peripheral and placental blood samples from pregnant women in Colombia. PLoS One. 2018 Aug 2;13(8):e0201769. doi: 10.1371/journal.pone.0201769. eCollection 2018. PMID 30071004
- [Derived] Tahita MC, Sondo P, Kabore B, Ilboudo H, Rouamba T, Sanou H, Ouedraogo K, Compaore A, Lompo P, Ouedraogo F, Sawadogo S, Derra K, Sawadogo YE, Some AM, Nana M, Sorgho H, Traore-Coulibaly M, Bassat Q, Tinto H. Impact and operational feasibility of adding malaria infection screening using an ultrasensitive RDT for placental and fetal outcomes in an area of high IPTP-SP coverage in Burkina Faso: the ASSER MALARIA pilot study protocol. Pilot Feasibility Stud. 2022 Oct 1;8(1):221. doi: 10.1186/s40814-022-01181-2. PMID 36183100